CLINICAL TRIAL: NCT00999544
Title: New Neural Drug Targets: An Evaluation of the Effects of Aprepitant on the Response to Oxycodone
Brief Title: Aprepitant Effects on Oxycodone Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sharon Walsh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Sharon Walsh, Director Center on Drug and Alcohol Research, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 09-0446; R01DA027031 (NIH)
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Results first posted 2013-08-23 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Narcotic Abuse
Keywords: opioid; oxycodone; NK1 antagonist; aprepitant; intranasal; abuse
MeSH Terms: conditions — Narcotic-Related Disorders | interventions — Aprepitant; Oxycodone

STUDY DESIGN:
Intervention Model Description: Within subject crossover designed that examined 15 experimental conditions within a single group of participants
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (15):
- Placebo aprepitant/0 mg oxycodone IN PO (Experimental): Placebo aprepitant/Placebo oxycodone IN/PO
  Interventions: Drug: Aprepitant 0mg; Drug: Oxycodone 0mg, p.o.; Drug: Oxycodone 0mg, IN
- Placebo aprepitant/ oxycodone 15 IN 0 PO (Experimental): Placebo aprepitant/ oxycodone 15 IN 0 PO
  Interventions: Drug: Aprepitant 0mg; Drug: Oxycodone 0mg, p.o.; Drug: Oxycodone 15mg, IN
- Placebo aprepitant/ oxycodone 30 IN 0 PO (Experimental): Placebo aprepitant/ oxycodone 30 IN 0 PO
  Interventions: Drug: Aprepitant 0mg; Drug: Oxycodone 0mg, p.o.; Drug: Oxycodone 30mg, IN
- Placebo aprepitant/ oxycodone 0 IN 20 PO (Experimental): Placebo aprepitant/ oxycodone 0 IN 20 PO
  Interventions: Drug: Aprepitant 0mg; Drug: Oxycodone 20mg, p.o.; Drug: Oxycodone 0mg, IN
- Placebo aprepitant/ oxycodone 0 IN 40 PO (Experimental): Placebo aprepitant/ oxycodone 0 IN 40 PO
  Interventions: Drug: Aprepitant 0mg; Drug: Oxycodone 40mg, p.o.; Drug: Oxycodone 0mg, IN
- Aprepitant 40 mg/ oxycodone 0 IN 0 PO (Experimental): Aprepitant 40 mg/ oxycodone 0 IN 0 PO
  Interventions: Drug: Aprepitant 40mg; Drug: Oxycodone 0mg, p.o.; Drug: Oxycodone 0mg, IN
- Aprepitant 40 mg/ oxycodone 0 IN 20 PO (Experimental): Aprepitant 40 mg/ oxycodone 0 IN 20 PO
  Interventions: Drug: Aprepitant 40mg; Drug: Oxycodone 20mg, p.o.; Drug: Oxycodone 0mg, IN
- Aprepitant 40 mg/ oxycodone 0 IN 40 PO (Experimental): Aprepitant 40 mg/ oxycodone 0 IN 40 PO
  Interventions: Drug: Aprepitant 40mg; Drug: Oxycodone 40mg, p.o.; Drug: Oxycodone 0mg, IN
- Aprepitant 40 mg/ oxycodone 15 IN 0 PO (Experimental): Aprepitant 40 mg/ oxycodone 15 IN 0 PO
  Interventions: Drug: Aprepitant 40mg; Drug: Oxycodone 0mg, p.o.; Drug: Oxycodone 15mg, IN
- Aprepitant 40 mg/ oxycodone 30 IN 0 PO (Experimental): Aprepitant 40 mg/ oxycodone 30 IN 0 PO
  Interventions: Drug: Aprepitant 40mg; Drug: Oxycodone 0mg, p.o.; Drug: Oxycodone 30mg, IN
- Aprepitant 200 mg/ oxycodone 0 IN 0 PO (Experimental): Aprepitant 200 mg/ oxycodone 0 IN 0 PO
  Interventions: Drug: Aprepitant 200mg; Drug: Oxycodone 0mg, p.o.; Drug: Oxycodone 0mg, IN
- Aprepitant 200 mg/ oxycodone 0 IN 20 PO (Experimental): Aprepitant 200 mg/ oxycodone 0 IN 20 PO
  Interventions: Drug: Aprepitant 200mg; Drug: Oxycodone 20mg, p.o.; Drug: Oxycodone 0mg, IN
- Aprepitant 200 mg/ oxycodone 0 IN 40 PO (Experimental): Aprepitant 200 mg/ oxycodone 0 IN 40 PO
  Interventions: Drug: Aprepitant 200mg; Drug: Oxycodone 40mg, p.o.; Drug: Oxycodone 0mg, IN
- Aprepitant 200 mg/ oxycodone 15 IN 0 PO (Experimental): Aprepitant 200 mg/ oxycodone 15 IN 0 PO
  Interventions: Drug: Aprepitant 200mg; Drug: Oxycodone 0mg, p.o.; Drug: Oxycodone 15mg, IN
- Aprepitant 200 mg/ oxycodone 30 IN 0 PO (Experimental): Aprepitant 200 mg/ oxycodone 30 IN 0 PO
  Interventions: Drug: Aprepitant 200mg; Drug: Oxycodone 0mg, p.o.; Drug: Oxycodone 30mg, IN

INTERVENTIONS:
Drug: Aprepitant 0mg — Aprepitant 0mg, p.o. pretreatment
  Arms: Placebo aprepitant/ oxycodone 0 IN 20 PO; Placebo aprepitant/ oxycodone 0 IN 40 PO; Placebo aprepitant/ oxycodone 15 IN 0 PO; Placebo aprepitant/ oxycodone 30 IN 0 PO; Placebo aprepitant/0 mg oxycodone IN PO
Drug: Aprepitant 40mg — Aprepitant 40mg, p.o. pretreatment
  Arms: Aprepitant 40 mg/ oxycodone 0 IN 0 PO; Aprepitant 40 mg/ oxycodone 0 IN 20 PO; Aprepitant 40 mg/ oxycodone 0 IN 40 PO; Aprepitant 40 mg/ oxycodone 15 IN 0 PO; Aprepitant 40 mg/ oxycodone 30 IN 0 PO
Drug: Aprepitant 200mg — Aprepitant 200mg, p.o. pretreatment
  Arms: Aprepitant 200 mg/ oxycodone 0 IN 0 PO; Aprepitant 200 mg/ oxycodone 0 IN 20 PO; Aprepitant 200 mg/ oxycodone 0 IN 40 PO; Aprepitant 200 mg/ oxycodone 15 IN 0 PO; Aprepitant 200 mg/ oxycodone 30 IN 0 PO
Drug: Oxycodone 0mg, p.o. — Oxycodone 0mg, p.o.
  Arms: Aprepitant 200 mg/ oxycodone 0 IN 0 PO; Aprepitant 200 mg/ oxycodone 15 IN 0 PO; Aprepitant 200 mg/ oxycodone 30 IN 0 PO; Aprepitant 40 mg/ oxycodone 0 IN 0 PO; Aprepitant 40 mg/ oxycodone 15 IN 0 PO; Aprepitant 40 mg/ oxycodone 30 IN 0 PO; Placebo aprepitant/ oxycodone 15 IN 0 PO; Placebo aprepitant/ oxycodone 30 IN 0 PO; Placebo aprepitant/0 mg oxycodone IN PO
Drug: Oxycodone 20mg, p.o. — Oxycodone 20mg, p.o.
  Arms: Aprepitant 200 mg/ oxycodone 0 IN 20 PO; Aprepitant 40 mg/ oxycodone 0 IN 20 PO; Placebo aprepitant/ oxycodone 0 IN 20 PO
Drug: Oxycodone 40mg, p.o. — Oxycodone 40mg, p.o.
  Arms: Aprepitant 200 mg/ oxycodone 0 IN 40 PO; Aprepitant 40 mg/ oxycodone 0 IN 40 PO; Placebo aprepitant/ oxycodone 0 IN 40 PO
Drug: Oxycodone 0mg, IN — Oxycodone 0mg, IN
  Arms: Aprepitant 200 mg/ oxycodone 0 IN 0 PO; Aprepitant 200 mg/ oxycodone 0 IN 20 PO; Aprepitant 200 mg/ oxycodone 0 IN 40 PO; Aprepitant 40 mg/ oxycodone 0 IN 0 PO; Aprepitant 40 mg/ oxycodone 0 IN 20 PO; Aprepitant 40 mg/ oxycodone 0 IN 40 PO; Placebo aprepitant/ oxycodone 0 IN 20 PO; Placebo aprepitant/ oxycodone 0 IN 40 PO; Placebo aprepitant/0 mg oxycodone IN PO
Drug: Oxycodone 15mg, IN — Oxycodone 15mg, IN
  Arms: Aprepitant 200 mg/ oxycodone 15 IN 0 PO; Aprepitant 40 mg/ oxycodone 15 IN 0 PO; Placebo aprepitant/ oxycodone 15 IN 0 PO
Drug: Oxycodone 30mg, IN — Oxycodone 30mg, IN
  Arms: Aprepitant 200 mg/ oxycodone 30 IN 0 PO; Aprepitant 40 mg/ oxycodone 30 IN 0 PO; Placebo aprepitant/ oxycodone 30 IN 0 PO

SUMMARY:
Addressing the issue of opioid dependence and tolerance has public health implications for the treatment of opioid abuse (both heroin as well as pharmaceutical opioids) and for the treatment of pain. Recent preclinical data suggest a role for Substance P (NK-1) receptors in modulating both the acute and chronic response to opioids. The objective of this study is to determine whether pretreatment with aprepitant, a selective neurokinin-1 (NK-1) antagonist can reduce the direct response to an opioid agonist (oxycodone) on measures related to abuse liability and reinforcing effects.

DETAILED DESCRIPTION:
Healthy adult volunteers with histories of illicit opioid use by the intranasal and oral routes will be admitted to this 6-week inpatient, crossover study. They will participate in 15 experimental test sessions, each lasting approximately 6.5 hours, during which they will receive a range of acute doses of aprepitant, including placebo, followed by challenge with oxycodone or placebo (given intranasally or orally). Multi-dimensional outcomes, including physiological (blood pressure, oxygen saturation, pupil diameter), subjective (questionnaires related to mood, abuse liability) and observer ratings will be collected repeatedly throughout each session. Data will be analyzed using parametric approaches to within-subject designs.

ELIGIBILITY:
Inclusion Criteria:

* Recreational user of opioids
* Healthy
* Ages 18-55 years old
* Able to provide informed consent

Exclusion Criteria:

* Ongoing medical or psychiatric condition that would be contraindicated for participation
* Past 30 day use of and P4503A4 inhibitor

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2009-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Walsh, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

REFERENCES:
- [Result] Walsh SL, Heilig M, Nuzzo PA, Henderson P, Lofwall MR. Effects of the NK1 antagonist, aprepitant, on response to oral and intranasal oxycodone in prescription opioid abusers. Addict Biol. 2013 Mar;18(2):332-43. doi: 10.1111/j.1369-1600.2011.00419.x. Epub 2012 Jan 19. PMID 22260216

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All recruitment was conducted through a research clinic at a public university.
Pre-assignment Details: Subjects were initially screened for inclusion/exclusion criteria. Fifteen subjects signed the screening consent but only nine were qualified to participate and signed the study consent. One subject left the study before receiving any interventions.
Groups:
- Within-subject Crossover Design: All subjects received exposure to every study condition in random order. During each of 15 separate test sessions, subjects received pretreatment with aprepitant (0, 40 or 200 mg) followed by a single challenge with a oxycodone (15 or 30, intranasal; 20 or 40 mg) or placebo. The fifteen dose conditions were administered in random order and each subject was exposed to each dose combination once.
Period: Overall Study
Arm/Group | Within-subject Crossover Design
Started | 9
Completed | 8
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Crossover Within Subject: All subjects were exposed to every condition.
Arm/Group | Crossover Within Subject
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Abuse Liability Proxy
Description: Visual analog scale ratings (from 0-100) on the subject-rated measure of "How much do you like the drug?" with higher scores indicating greater abuse liability (and 100 anchored with "extremely" and zero indicating none anchored with "none at all." Data were collected across multiple time points but the peak maximum score was used for the primary outcome measure.
Time Frame: 42 days
Population: Prior laboratory-based within subject studies of the pharmacodynamic response to opioid challenges. The within subject data analysis does not lend itself to reporting data in the format provided below.
Measure: Mean (Standard Deviation); unit: units on a scale (points 0-100)
Groups:
- Placebo-Placebo (in and po); Aprepitant 40 mg - Placebo; Aprepitant 200 mg- Placebo; Placebo- 15 mg Oxycodone Intranasal; Placebo- 30 mg Oxycodone Intranasal; Placebo- 20 mg Oxycodone Oral; Placebo - 40 mg Oxycodone Oral; Aprepitant 40 mg- 15 mg Oxycodone Intranasal; Aprepitant 40 mg - 30 mg Oxycodone Intranasal; Aprepitant 40 mg- 20 mg Oxycodone Oral; Aprepitant 40 mg - 40 mg Oxycodone Oral; Aprepitant 200 mg - 15 mg Oxycodone Intranasal; Aprepitant 200 mg - 30 mg Oxycodone Intranasal; Aprepitant 200 mg- 20 Oxycodone Oral; Aprepitant 200 mg- 40 Oxycodone Oral: All subjects received exposure to this study condition once.
Arm/Group | Placebo-Placebo (in and po) | Aprepitant 40 mg - Placebo | Aprepitant 200 mg- Placebo | Placebo- 15 mg Oxycodone Intranasal | Placebo- 30 mg Oxycodone Intranasal | Placebo- 20 mg Oxycodone Oral | Placebo - 40 mg Oxycodone Oral | Aprepitant 40 mg- 15 mg Oxycodone Intranasal | Aprepitant 40 mg - 30 mg Oxycodone Intranasal | Aprepitant 40 mg- 20 mg Oxycodone Oral | Aprepitant 40 mg - 40 mg Oxycodone Oral | Aprepitant 200 mg - 15 mg Oxycodone Intranasal | Aprepitant 200 mg - 30 mg Oxycodone Intranasal | Aprepitant 200 mg- 20 Oxycodone Oral | Aprepitant 200 mg- 40 Oxycodone Oral
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
units on a scale (points 0-100) | 0.197 (0.197) | 0.483 (0.397) | 0.159 (0.159) | 7.678 (2.656) | 17.450 (4.275) | 9.850 (5.090) | 16.646 (4.203) | 8.543 (2.892) | 15.092 (4.706) | 13.281 (4.009) | 17.244 (4.788) | 17.195 (4.897) | 28.211 (4.365) | 8.196 (2.667) | 26.322 (3.702)
Statistical Analysis 1: Comparison: Placebo-Placebo (in and po) vs Aprepitant 40 mg - Placebo vs Aprepitant 200 mg- Placebo vs Placebo- 15 mg Oxycodone Intranasal vs Placebo- 30 mg Oxycodone Intranasal vs Placebo- 20 mg Oxycodone Oral vs Placebo - 40 mg Oxycodone Oral vs Aprepitant 40 mg- 15 mg Oxycodone Intranasal vs Aprepitant 40 mg - 30 mg Oxycodone Intranasal vs Aprepitant 40 mg- 20 mg Oxycodone Oral vs Aprepitant 40 mg - 40 mg Oxycodone Oral vs Aprepitant 200 mg - 15 mg Oxycodone Intranasal vs Aprepitant 200 mg - 30 mg Oxycodone Intranasal vs Aprepitant 200 mg- 20 Oxycodone Oral vs Aprepitant 200 mg- 40 Oxycodone Oral; Area-under-the-curve (AUC) scores were derived from time course data and analyzed using two-factor ANOVA [aprepitant dose (3 levels)x oxycodone dose (3 levels)]. All analyses were conducted using SAS 9.1 for Windows (SAS Institute Inc., Cary, NC, USA) and were considered significant when P 0.05; Test type: Superiority or Other; p < .05, ANOVA

2. Secondary Outcome: Respiration Depression
Description: Respiration rate measured over 60 seconds. Data were collected across multiple time points, but the peak minimum score was used for this outcome measure.
Time Frame: 42 days
Population: Prior laboratory-based within subject studies of the pharmacodynamic response to opioid challenges.
Measure: Mean (Standard Deviation); unit: number of breaths per minute
Arm/Group | Placebo Aprepitant/0 mg Oxycodone IN PO | Placebo Aprepitant/ Oxycodone 15 IN 0 PO | Placebo Aprepitant/ Oxycodone 30 IN 0 PO | Placebo Aprepitant/ Oxycodone 0 IN 20 PO | Placebo Aprepitant/ Oxycodone 0 IN 40 PO | Aprepitant 40 mg/ Oxycodone 0 IN 0 PO | Aprepitant 40 mg/ Oxycodone 0 IN 20 PO | Aprepitant 40 mg/ Oxycodone 0 IN 40 PO | Aprepitant 40 mg/ Oxycodone 15 IN 0 PO | Aprepitant 40 mg/ Oxycodone 30 IN 0 PO | Aprepitant 200 mg/ Oxycodone 0 IN 0 PO | Aprepitant 200 mg/ Oxycodone 0 IN 20 PO | Aprepitant 200 mg/ Oxycodone 0 IN 40 PO | Aprepitant 200 mg/ Oxycodone 15 IN 0 PO | Aprepitant 200 mg/ Oxycodone 30 IN 0 PO
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
number of breaths per minute | 13.75 (3.15) | 11.63 (1.60) | 11.25 (1.75) | 12.13 (2.30) | 10.25 (1.98) | 12.25 (2.19) | 12.25 (2.12) | 11.00 (2.33) | 12.38 (1.92) | 11.63 (2.56) | 14.00 (2.33) | 14.00 (2.33) | 12.13 (2.17) | 12.00 (1.93) | 11.38 (3.02)

ADVERSE EVENTS:
Groups:
- Within-subject Crossover Design: All subjects received exposure to every study condition in random order. This was not a parallel group design.
Arm/Group | Within-subject Crossover Design
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
No significant adverse effects occurred. No adverse events led to study drop-out.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No